CLINICAL TRIAL: NCT02491086
Title: Motivating Smokers at Outdoor Public Smoking Hotspots to Have Quit Attempt With Nicotine Replacement Therapy Sampling: A Randomized Controlled Trial
Brief Title: Motivating Smokers at Outdoor Public Smoking Hotspots to Have Quit Attempt With Nicotine Replacement Therapy Sampling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Derek Yee-Tak Cheung, Post-doctoral Fellow, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201409176211
Record Dates: First submitted 2015-07-02; First posted 2015-07-07 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Smoking Cessation
Keywords: intervention, nicotine replacement sampling, smoking cessation, smoking hotspots
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive a free pack of one-week NRT. The nurse will help the subject to decide which NRT product (patch, gum and lozenge) he/she can use and advise how to use the NRT based on his/her smoking habit and amount of cigarette consumption, followed by the delivery of the sampling, instructions of using the NRT sampling, an education card about NRT and a 12-page smoking cessation booklet (Figure 1). Based on the experience in the previous trials, the choice of NRT (either patch, lozenge or gum) will be made according to subject's preference, and the counsellors will provide medication counselling [25-27]. If the subject is willing to continue the counselling at recruitment, the ambassador will further introduce the NRT's side effects, adherence and effectiveness (Table 1). Otherwise, the ambassador will contact the subject for providing these details and enquiring the usage through telephone within 2 days.
  Interventions: Drug: Nicotine replacement therapy (NRT) sampling; Behavioral: Smoking cessation counseling
- Control (Active Comparator): The control group subjects will only be advised by the ambassador to purchase the NRT on their own, but will not be given the sampling. The same education card and the 12-page smoking cessation booklet will be provided.
  Interventions: Behavioral: Smoking cessation counseling

INTERVENTIONS:
Drug: Nicotine replacement therapy (NRT) sampling — 1-week free NRT
  Arms: Intervention
Behavioral: Smoking cessation counseling — Smoking cessation counseling

SUMMARY:
Background About half of the daily smokers in Hong Kong have never tried and have no intention to quit smoking. 37.9% of daily smokers attempted to quit but failed. Nicotine replacement therapy (NRT) is a safe and effective pharmacotherapy to reduce withdrawal symptoms during early stage of tobacco abstinence and increase quit rate. However, the prevalence of using NRT in Hong Kong is lower than most of the developed countries. The proposed project aims to test if providing free NRT sampling to smokers can increase quit attempt and hence quit successfully.

Methods Nurses and university undergraduate students will be trained, and will invite smokers at outdoor public places to participate in the randomized controlled trial, which randomized eligible smokers to intervention or control group. The intervention group will be provided with 1-week free NRT sampling and medication counselling, whereas the control group will only be advised to purchase NRT on their own. The primary outcome is the proportion of any self-reported quit attempt (no smoking for at least 24 hours) in the past month at 1- and 3-month telephone follow-up.

Discussions The findings will inform the feasibility and effectiveness of delivering free NRT sampling to increase quit attempt and abstinence. It will yield more information on smokers' adherence to the NRT sampling, side effect and safety issue of the usage. Moreover, it will guide a future larger trial to test the effect from the NRT sampling and translation to practice.

DETAILED DESCRIPTION:
Trial design The study aims at motivating smokers to have quit attempt using nicotine replacement therapy (NRT) sampling. We will firstly train nurses and university undergraduate students as outreach smoking cessation ambassadors. These trained ambassadors will proactively approach the smokers at outdoor smoking hotspots, where rubbish bins with a collector of cigarette butts are nearby, and invite them to participate in the RCT.

Subjects Smokers with the following inclusion criteria will be invited to participate in our RCT: (1) Aged 18 years or above; (2) Smoke 10 cigarettes or more per day in the past week; (3) Able to read and speak Chinese; (4) Have not used NRT for the past 3 months; (5) Have no severe angina and serious cardiac arrhythmias; (6) Have not suffered from acute myocardial event in the past 4 weeks; and (7) Not pregnant and breastfeeding The recruitments of subjects will take place at 9 outdoor urban places where smokers stayed and smoked from July 2015 to September 2015 (To be confirmed) Procedures We target to train nurses and smoking cessation ambassadors for the recruitment and providing intervention to the subjects. Recruitment of outreach smoking cessation ambassadors will be conducted through sending mass mails to students of the University of Hong Kong. Retired nurses who are now providing counselling services in our existing smoking cessation projects will be recruited. They will be invited to participate in a training programme which provides them an overview of the smoking cessation counselling and pharmacotherapy in helping smokers quit smoking. Our research team (comprised of physicians and nurses) will develop the training material and intervention guide based on the principles of the US Agency for Health Care Policy and Research (AHCPR) guidelines in the US [28], the guidelines of the National Institutes of Health [29] and World Health Organization [30]. The training content will cover (1) smoking trend in Hong Kong; (2) health hazards of smoking, (3) basic skills in assessing smoking dependence and quitting readiness; (4) knowledge of smoking cessation medication (types of NRT, adherence and side effects etc.) and (5) brief counseling skills. At the end of the training, participants should be capable of delivering brief intervention of smoking cessation including the advice on using NRT.

Smoking cessation ambassadors will approach the smokers and distribute souvenirs with smoking cessation messages at the outdoor smoking hotspots. The souvenir will be a small pack of tissue paper, with motivational messages (e.g. 1 in 2 smokers will be killed by smoking), quitline number (e.g. Quitline of Tobacco Control Office 1833183) and other resources for quitting printed on the tissue pack. If the smoker is willing to accept the souvenir and talk to the ambassador, the ambassador will ask further questions related to the eligibility through an informal conversation. If the subject is eligible, the ambassador will seek his/her consent to receive further intervention and provide his/her mobile phone number.

Interventions The intervention group will receive a free pack of one-week NRT. The nurse will help the subject to decide which NRT product (patch, gum and lozenge) he/she can use and advise how to use the NRT based on his/her smoking habit and amount of cigarette consumption, followed by the delivery of the sampling, instructions of using the NRT sampling, an education card about NRT and a 12-page smoking cessation booklet (Figure 1). Based on the experience in the previous trials, the choice of NRT (either patch, lozenge or gum) will be made according to subject's preference, and the counsellors will provide medication counselling [25-27]. If the subject is willing to continue the counselling at recruitment, the ambassador will further introduce the NRT's side effects, adherence and effectiveness (Table 1). Otherwise, the ambassador will contact the subject for providing these details and enquiring the usage through telephone within 2 days.

Some subjects may not be interested to use NRT sampling or some may not use them for quitting it. An envelope with a return address and pre-paid postage will be given with the NRT sampling, so that subjects can send back any unused NRT sampling to us to avoid wastage.

The control group subjects will only be advised by the ambassador to purchase the NRT on their own, but will not be given the sampling. The same education card and the 12-page smoking cessation booklet will be provided.

Outcomes The primary outcome of the RCT is the proportion of any self-reported quit attempt (no smoking for at least 24 hours) in the past month at the 1- and 3-month follow-up. The secondary outcomes are (1) self-reported 7-day point prevalence of abstinence at 1-, 3- and 6-month follow-up; (2) perceived importance, confidence and difficulty to quit (scale 0-10) at all the follow-ups; (3) proportion of using all free NRT samples; (4) biochemically validated abstinence at 1-month follow-up.

At 1 week, 1, 3 and 6 months after the recruitment, all subjects will be contacted by a trained interviewer via telephone to assess their smoking status and discuss any difficulties they might have encountered. At least 7 call attempts at different time will be made before the subject is considered as loss to follow-up. Subjects who report no smoking in the past 7 days will be considered as self-reported quitters. Self-reported quitters at 1 month will be invited to participate in a biochemical validation including measurement of exhaled carbon monoxide (CO) and salivary cotinine level by NicAlert® strips (www.nymox.com). The criteria for validated abstinence were exhaled CO < 4 ppm and salivary cotinine < 10ng/ml [31, 32].

Sample size determination Since the RCT will test the feasibility and generate preliminary estimates of effectiveness of the NRT sampling, we propose the sample size as 50 for each arm (i.e. total sample size = 100). A similar RCT conducted by Jardin et al. (2014) which evaluated the effectiveness of 2-week free NRT to help non-motivated smokers to quit smoking was chosen for the power estimation. The results showed that the 3-month quit attempt rate of receiving free NRT was significantly higher than those who only received a quitline referral only (32% vs 16%, p=0.05). The relative risk (RR) is therefore determined (32%/16% = 2.0). Based on the RR of 2.0, and the 100 subjects, the power and type I error for detecting the difference using the Fisher's exact test will be 69.7% and 0.08.

Randomization Sequentially numbered, opaque sealed envelopes (SNOSE) and block randomization will be used to allocate subjects into two RCT groups. The primary investigator will prepare 100 identical, opaque, sealed, A5-sized envelops. 50 of them will each contain an eligibility form, an education card of NRT, an action plan for the intervention group, and an empty box of NRT. The other 50 envelops will contain the same eligibility form and education card, and an action plan for the control group. The ambassador will create a block of 4 envelops, with 2 in the intervention group and 2 in the control, and shuffle them thoroughly and contain them in a separate pile. Recruitment staff will use 1 of the 25 piles of the envelopes and randomly select 1 envelope for the intervention.

Allocation concealment The group allocations were concealed to the subjects and the ambassador. Subjects will not be aware of the allocation throughout the study.

Blinding As the assessors of the outcomes will be blinded to the group allocation, this RCT will be single-blinded.

Data analyses All data will be entered and analyzed with SPSS for Windows version 20. The rate of quit attempt and 7-day abstinence will be assessed with t-test and odds ratio from logistic regression. Both intention-to-treat (assuming missing subjects have no changes) and complete case analysis will be done.

Ethics NRT for smoking cessation was proved as an effective and safe aid to smoking cessation, which can be purchased over-the-counter in pharmacy or freely prescribed in the smoking cessation clinics in Hong Kong. Common side effect of nicotine patch is skin reaction. About 50% of patients using the nicotine patch will experience a local skin reaction. The reaction is usually mild and self-limiting, but occasionally worsens over the course of therapy. Local treatment with hydrocortisone cream (1%) or triamcinolone cream (0.5%) and rotating patch sites may ameliorate such local reaction. In fewer than 5% of patients, such reaction requires the discontinuation of the NRT. Other side effects are insomnia and/or vivid dreams. Common side effects of nicotine gum include mouth soreness, hiccups, dyspepsia, and jaw ache. These effects are generally mild and transient and often can be alleviated by correcting the patient's chewing technique. [10] These effects are generally mild and can be alleviated by correcting the patient's using habit. All subjects will be asked at the first 7-day telephone follow-up if they have the above side effects. If so, the counsellor will provide counselling on the usage. If the side effects are serious, counsellor will ask them to cease the usage and mail back the sampling.

ELIGIBILITY:
Inclusion criteria:

1. Aged 18 years or above;
2. Smoke 10 cigarettes or more per day in the past week;
3. Able to read and speak Chinese;
4. Have not used NRT for the past 3 months

Exclusion criteria:

1. Have severe angina and serious cardiac arrhythmias;
2. Have suffered from acute myocardial event in the past 4 weeks;
3. Pregnant and breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-07; Primary Completion 2016-01 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Self-reported quit attempt | 1 month
  No smoking for at least 24 hours in the past month

SECONDARY OUTCOMES:
Self-reported 7-day prevalence of tobacco abstinence | 1 month
Proportion of participants using NRT in the past month | 1 month
Biochemically validated quit rate, measurement of exhaled carbon monoxide | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Yee Tak Derek Cheung, Cheung, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] McGhee SM, Ho LM, Lapsley HM, Chau J, Cheung WL, Ho SY, Pow M, Lam TH, Hedley AJ. Cost of tobacco-related diseases, including passive smoking, in Hong Kong. Tob Control. 2006 Apr;15(2):125-30. doi: 10.1136/tc.2005.013292. PMID 16565461
- [Background] Koplan JP, An WK, Lam RM. Hong Kong: a model of successful tobacco control in China. Lancet. 2010 Apr 17;375(9723):1330-1. doi: 10.1016/S0140-6736(10)60398-4. Epub 2010 Mar 25. No abstract available. PMID 20347129
- [Background] Census & Statistics Department (Hong Kong SAR government): Thematic Household Survey, Report No. 53: Pattern of Smoking. In. Hong Kong: Census & Statistics Department; 2013
- [Background] Hong Kong Council on Smoking and Health: June 2013, COSH Report No. 16 - Quit to Win 2010 and smoking cessation. In. Hong Kong: Hong Kong Council on Smoking Health; 2013.
- [Background] Kasza KA, Hyland AJ, Borland R, McNeill AD, Bansal-Travers M, Fix BV, Hammond D, Fong GT, Cummings KM. Effectiveness of stop-smoking medications: findings from the International Tobacco Control (ITC) Four Country Survey. Addiction. 2013 Jan;108(1):193-202. doi: 10.1111/j.1360-0443.2012.04009.x. Epub 2012 Aug 14. PMID 22891869
- [Background] Lancaster T, Stead L, Silagy C, Sowden A. Effectiveness of interventions to help people stop smoking: findings from the Cochrane Library. BMJ. 2000 Aug 5;321(7257):355-8. doi: 10.1136/bmj.321.7257.355. No abstract available. PMID 10926597
- [Background] Song F, Raftery J, Aveyard P, Hyde C, Barton P, Woolacott N. Cost-effectiveness of pharmacological interventions for smoking cessation: a literature review and a decision analytic analysis. Med Decis Making. 2002 Sep-Oct;22(5 Suppl):S26-37. doi: 10.1177/027298902237708. PMID 12369228
- [Background] Borland R, Li L, Driezen P, Wilson N, Hammond D, Thompson ME, Fong GT, Mons U, Willemsen MC, McNeill A, Thrasher JF, Cummings KM. Cessation assistance reported by smokers in 15 countries participating in the International Tobacco Control (ITC) policy evaluation surveys. Addiction. 2012 Jan;107(1):197-205. doi: 10.1111/j.1360-0443.2011.03636.x. PMID 21883605
- [Background] 2008 PHS Guideline Update Panel, Liaisons, and Staff. Treating tobacco use and dependence: 2008 update U.S. Public Health Service Clinical Practice Guideline executive summary. Respir Care. 2008 Sep;53(9):1217-22. No abstract available. PMID 18807274
- [Background] National Institue for Clinical Excellence: Guidance on the use of nicotine replacement therapy (NRT) and bupropion for smoking cessation. In. NHS, London: National Institue for Clinical Excellence; 2002.
- [Background] Prochaska JO, Velicer WF. The transtheoretical model of health behavior change. Am J Health Promot. 1997 Sep-Oct;12(1):38-48. doi: 10.4278/0890-1171-12.1.38. PMID 10170434
- [Background] West R, Sohal T. "Catastrophic" pathways to smoking cessation: findings from national survey. BMJ. 2006 Feb 25;332(7539):458-60. doi: 10.1136/bmj.38723.573866.AE. Epub 2006 Jan 27. PMID 16443610
- [Background] Jimenez-Muro A, Nerin I, Samper P, Marqueta A, Beamonte A, Gargallo P, Oros D, Rodriguez G. A proactive smoking cessation intervention in postpartum women. Midwifery. 2013 Mar;29(3):240-5. doi: 10.1016/j.midw.2012.01.003. Epub 2012 Feb 22. PMID 22361008
- [Background] Carpenter MJ, Hughes JR, Gray KM, Wahlquist AE, Saladin ME, Alberg AJ. Nicotine therapy sampling to induce quit attempts among smokers unmotivated to quit: a randomized clinical trial. Arch Intern Med. 2011 Nov 28;171(21):1901-7. doi: 10.1001/archinternmed.2011.492. PMID 22123796
- [Background] Jardin BF, Cropsey KL, Wahlquist AE, Gray KM, Silvestri GA, Cummings KM, Carpenter MJ. Evaluating the effect of access to free medication to quit smoking: a clinical trial testing the role of motivation. Nicotine Tob Res. 2014 Jul;16(7):992-9. doi: 10.1093/ntr/ntu025. Epub 2014 Mar 7. PMID 24610399
- [Background] Larabie LC. To what extent do smokers plan quit attempts? Tob Control. 2005 Dec;14(6):425-8. doi: 10.1136/tc.2005.013615. PMID 16319368
- [Background] Ferguson SG, Shiffman S, Gitchell JG, Sembower MA, West R. Unplanned quit attempts--results from a U.S. sample of smokers and ex-smokers. Nicotine Tob Res. 2009 Jul;11(7):827-32. doi: 10.1093/ntr/ntp072. Epub 2009 Jun 9. PMID 19509277
- [Background] Murray RL, Lewis SA, Coleman T, Britton J, McNeill A. Unplanned attempts to quit smoking: missed opportunities for health promotion? Addiction. 2009 Nov;104(11):1901-9. doi: 10.1111/j.1360-0443.2009.02647.x. Epub 2009 Aug 4. PMID 19681806
- [Background] Shiffman S, Ferguson SG, Rohay J, Gitchell JG. Perceived safety and efficacy of nicotine replacement therapies among US smokers and ex-smokers: relationship with use and compliance. Addiction. 2008 Aug;103(8):1371-8. doi: 10.1111/j.1360-0443.2008.02268.x. PMID 18855827
- [Background] Ferguson SG, Gitchell JG, Shiffman S, Sembower MA, Rohay JM, Allen J. Providing accurate safety information may increase a smoker's willingness to use nicotine replacement therapy as part of a quit attempt. Addict Behav. 2011 Jul;36(7):713-6. doi: 10.1016/j.addbeh.2011.02.002. Epub 2011 Feb 13. PMID 21371825
- [Background] Vogt F, Hall S, Marteau TM. Understanding why smokers do not want to use nicotine dependence medications to stop smoking: qualitative and quantitative studies. Nicotine Tob Res. 2008 Aug;10(8):1405-13. doi: 10.1080/14622200802239280. PMID 18686189
- [Background] Lindson-Hawley N, Aveyard P, Hughes JR. Reduction versus abrupt cessation in smokers who want to quit. Cochrane Database Syst Rev. 2012 Nov 14;11:CD008033. doi: 10.1002/14651858.CD008033.pub3. PMID 23152252
- [Background] Asfar T, Ebbert JO, Klesges RC, Relyea GE. Do smoking reduction interventions promote cessation in smokers not ready to quit? Addict Behav. 2011 Jul;36(7):764-8. doi: 10.1016/j.addbeh.2011.02.003. Epub 2011 Feb 12. PMID 21420791
- [Background] A clinical practice guideline for treating tobacco use and dependence: A US Public Health Service report. The Tobacco Use and Dependence Clinical Practice Guideline Panel, Staff, and Consortium Representatives. JAMA. 2000 Jun 28;283(24):3244-54. PMID 10866874
- [Background] Medline Plus: Nicotine Replacement Therapy. In: Nicotine Replacement Therapy: MedlinePlus Medical Encyclopedia U.S.: U.S. National Library of Medicine, National Insititutes of Health; 2009.
- [Background] World Health Organization: Adherence to long-term therapies: Evidence for action. In. Geneva: World Health Organization; 2003.
- [Background] Abdullah AS, Hedley AJ, Chan SS, Lam TH. A randomized controlled trial of two different lengths of nicotine replacement therapy for smoking cessation. Biomed Res Int. 2013;2013:961751. doi: 10.1155/2013/961751. Epub 2013 Sep 9. PMID 24089693
- [Background] Chan SS, Leung DY, Abdullah AS, Wong VT, Hedley AJ, Lam TH. A randomized controlled trial of a smoking reduction plus nicotine replacement therapy intervention for smokers not willing to quit smoking. Addiction. 2011 Jun;106(6):1155-63. doi: 10.1111/j.1360-0443.2011.03363.x. Epub 2011 Mar 7. PMID 21226883
- [Background] Lam TH, Abdullah AS, Chan SS, Hedley AJ; Hong Kong Council on Smoking and Health Smoking Cessation Health Centre (SCHC) Steering Group. Adherence to nicotine replacement therapy versus quitting smoking among Chinese smokers: a preliminary investigation. Psychopharmacology (Berl). 2005 Feb;177(4):400-8. doi: 10.1007/s00213-004-1971-y. Epub 2004 Jul 29. PMID 15289997
- [Background] Cooke F, Bullen C, Whittaker R, McRobbie H, Chen MH, Walker N. Diagnostic accuracy of NicAlert cotinine test strips in saliva for verifying smoking status. Nicotine Tob Res. 2008 Apr;10(4):607-12. doi: 10.1080/14622200801978680. PMID 18418783
- [Background] Javors MA, Hatch JP, Lamb RJ. Cut-off levels for breath carbon monoxide as a marker for cigarette smoking. Addiction. 2005 Feb;100(2):159-67. doi: 10.1111/j.1360-0443.2004.00957.x. PMID 15679745
- [Background] Yang J, Hammond D, Driezen P, Fong GT, Jiang Y. Health knowledge and perception of risks among Chinese smokers and non-smokers: findings from the Wave 1 ITC China Survey. Tob Control. 2010 Oct;19 Suppl 2(Suppl 2):i18-23. doi: 10.1136/tc.2009.029710. PMID 20935195
- [Derived] Cheung YT, Leung JP, Cheung CK, Li WH, Wang MP, Lam TH. Motivating smokers at outdoor public smoking hotspots to have a quit attempt with a nicotine replacement therapy sample: study protocol for a randomized controlled trial. Trials. 2016 Jul 26;17(1):355. doi: 10.1186/s13063-016-1485-z. PMID 27456342